CLINICAL TRIAL: NCT03082625
Title: Topical Magnesium Supplementation for the Treatment of Muscle Cramps in Dialysis Patients
Brief Title: Topical Magnesium and Muscle Cramps in Dialysis Patients.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Charles Gairdner Hospital (Other)
Responsible Party: Principal Investigator, Neil Boudville, Head of Deparment of Renal Medicine, Sir Charles Gairdner Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-158
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease; Dialysis Related Complications
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: Randomised placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical delivery systems and appearance of the product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdermal Magnesium (Experimental): 5 sprays each on the 2 most effected areas for muscle cramps twice a day
  Interventions: Drug: Transdermal Magnesium
- Placebo (Placebo Comparator): 5 sprays each on the 2 most effected areas for muscle cramps twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Transdermal Magnesium — Magnesium
  Other Names: Topical Magnesium
  Arms: Transdermal Magnesium
Drug: Placebo
  Arms: Placebo

SUMMARY:
Oral magnesium supplementation has been widely used in the treatment of muscle cramps. Muscle cramps are common in dialysis patients but are not satisfactorily prevented by oral magnesium. Transdermal administration of magnesium has been promoted as a potential treatment for muscle cramps but this has not been investigated rigorously. We aim to evaluate the effectiveness of transdermal magnesium supplementation in reducing cramp frequency and severity. We will recruit current haemodialysis patients who suffer from muscle cramps into a randomised, placebo-controlled, cross-over design trial. Each intervention period will last 8 weeks with a 4-week washout period in between. We will measure muscle cramp frequency, duration and severity as the primary outcomes.

DETAILED DESCRIPTION:
Study participants will be provided with a cramp diary in which they will record the date, time, duration and severity of any muscle cramps they experience. Severity will be measured using a Likert scale in which participants will be asked to mark along a 10 cm line the severity of the pain they have experienced with each muscle cramp (ranging from no pain to the worst pain possible). The distance between "no pain" and the participant's mark will then be measured in centimetres (to one decimal point) to provide a precise value for muscle cramp severity. Participants will also be asked to record the duration of each muscle cramp they experience to the nearest minute.

Patients will be asked to record in their cramp diaries the nature of any unwanted skin changes they may have experienced during their participation in the study including when they first noticed these changes and the duration in which they were affected by them.

Serum magnesium, calcium and potassium levels will be measured and recorded before commencement of the study, at the end of the first stage of the study, at the end of the washout out period and at the end of the second stage of the study.

Patients will also be asked to describe their restless leg symptoms at different periods of the study from - no different to usual, better, much better, worse, much worse.

Participants will be seen by the investigators at enrolment into the study and at the end of the run-in period, first treatment period and second treatment period. In addition, participants will be asked to fill in a Likert scale regarding their views on how effective they believe the treatments were after each treatment period.

5.2 Study Plan

During the run-in period patients will make no changes to their treatments for their muscle cramps. During the treatment periods patients will be asked to apply five sprays of the intervention or placebo to the two sites of the body most commonly affected by muscle cramps, twice daily. During the two-week wash-out period there will be no spray applied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic kidney disease and receiving dialysis treatment
* Previous experience of at least 2 or more muscle cramps per month in at least 3 of the last 6 months
* Men or women aged 18 years and older
* Capacity to provide informed consent

Exclusion Criteria:

* Patients less than 18 years of age
* Women who are pregnant and the human fetus
* Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study and/or likely to cause death within the study duration
* Participation in another clinical during the last 12 weeks
* Known allergic reactions against any component of the study drug or its comparator(s)
* Known contraindication to any component of the study drug or its comparator(s)
* Concurrent diseases which exclude the administration of therapy as outlined by the study protocol
* Subjects who, in the opinion of the investigator, are not likely to complete the study for whatever reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the average number of muscle cramps per week between magnesium and placebo treatments | 3 weeks
  final 3 weeks

SECONDARY OUTCOMES:
Difference in average cramp duration between magnesium and placebo treatments | 3 weeks
  final 3 weeks
Difference in average cramp severity between magnesium and placebo treatments | 3 weeks
  final 3 weeks
Percentage change in serum magnesium concentration from baseline and at the end of each treatment stage | 3 weeks
Difference in restless legs symptoms between the magnesium and placebo treatment stages. | 3 weeks

IPD SHARING:
Plan to Share IPD: Undecided
The plan at this stage is to have unidentified information available in a secure web-based environment.

REFERENCES:
- [Derived] Garrison SR, Korownyk CS, Kolber MR, Allan GM, Musini VM, Sekhon RK, Dugre N. Magnesium for skeletal muscle cramps. Cochrane Database Syst Rev. 2020 Sep 21;9(9):CD009402. doi: 10.1002/14651858.CD009402.pub3. PMID 32956536